CLINICAL TRIAL: NCT04982120
Title: A Post-510(k) Study of Patients With Overactive Bladder (OAB) Treated With OnabotulinumtoxinA (Botox, Allergan PLC) Using the Repris Bladder Injection System
Brief Title: Use of Repris Needle in Bladder Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uro-1 Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Repris Botox Study
Record Dates: First submitted 2021-07-15; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Repris Needle (Experimental): Reprise sheath and needle
  Interventions: Device: Repris Needle

INTERVENTIONS:
Device: Repris Needle — Injection of Botox

SUMMARY:
Treatment of overactive bladder (OAB) has been treated successfully by the injection of Botox. The Repris injection needle has a deflection that may assist in injection difficult to reach with standard straight needles. This study will assess the success, safety and patient tolerance of this new injection needle.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm study of the Repris injection needle to administer Botox to the bladder wall in patients with an overactive bladder. Following advancement of a cystoscope to the patient's bladder, the Repris needle will be advanced to the area of interest and into the bladder wall in order to administer the recommended volume of Botox. After injection, the needle will be removed and the procedure will be concluded. The patient will be asked to rank her tolerance of the procedure and level of discomfort using a standardized pain scale before being released. Five days after the procedure the patient will be contacted by telephone to determine whether any adverse events had occurred since release.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Able to undergo routine cystoscopy
* Willing to provide verbal assessment of her condition within 5 days after the procedure

Exclusion Criteria:

* History of urethral strictures
* Presence of a suprapubic catheter or tube due to urethral trauma
* history of interstitial cystitis
* currently being treated for a urinary tract infection (UTI)
* gross hematuria present
* Known allergy or sensitivity to any component of the medication or solution to be injected during the study
* is pregnant, lactating, or with child-bearing potential unable or unwilling to use a reliable form of contraception while participating in the study
* cannot empty her bladder on her own and is routinely catheterizing the urethra
* unable to read, understand, and/or provide a ranking of pain level during the procedure,
* unable or unwilling to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Overactive bladder syndrome is more frequently treated in females than males
Enrollment: 40 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-07-14 (Estimated)

PRIMARY OUTCOMES:
Procedure Success | 1 Day of the procedure
  Percentage of subjects with successful injection of medication

SECONDARY OUTCOMES:
Patient Tolerance of Injection | 1 Day of the procedure
  Level of pain from use of the needle measured on Likert Scale 1 to 5
Adverse Events during Procedure | Day 0 and Day 5
  Incidence and Severity of Adverse events associated with the injection

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lawson, PhD, Study Director — Uro-1 Medical
Locations (1):
- Georgia Urology, Cartersville, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient identification will not be shared
Supporting Information: Study Protocol, ICF
Time Frame: Within 7 days after completion of study
Access Criteria: Permission from PI